CLINICAL TRIAL: NCT00658073
Title: Autologous Bone Marrow Mesenchymal Stem Cell Transplantation in Recipients of Living Kidney Allografts
Brief Title: Induction Therapy With Autologous Mesenchymal Stem Cells for Kidney Allografts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: Jianming Tan M.D and Ph.D, Fuzhou General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSC-K-2
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-02

CONDITIONS: Renal Transplant Rejection
Keywords: Kidney transplant; Mesenchymal stem cell (MSC)
MeSH Terms: interventions — Kidney Transplantation; cni protein, Drosophila

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Active Comparator): Patients in Group A will receive MSCs instead of anti-interleukin 2 receptor antibody for induction therapy. The first MSCs infusion intravenously will be right at releasing renal artery clamp to establish allograft blood flow and the second infusion of MSCs will be performed two weeks after transplantation. Patients will receive standard regular immunosuppressive agents including calcineurin inhibitor, glucocorticoid, and MMF.
  Interventions: Procedure: Kidney transplantation with MSCs infusion
- B (Active Comparator): Patients in Group B will receive MSCs instead of anti-interleukin 2 receptor antibody for induction therapy. The first MSCs infusion intravenously will be right at releasing renal artery clamp to establish allograft blood flow and the second infusion of MSCs will be performed two weeks after transplantation. Patients will receive 80% less of calcineurin inhibitor than in Group A. Other immunosuppressive agents such as glucocorticoid and MMF remained the same doses as in Group A.
  Interventions: Procedure: Kidney transplantation with MSCs infusion
- C (Active Comparator): Patients in Group C will receive anti-interleukin 2 receptor antibody (Basiliximab)for induction therapy. Patients will receive the same doses of regular immunosuppressive agents including calcineurin inhibitor, glucocorticoid, and MMF as in Group A.
  Interventions: Procedure: kidney transplantation without MSC infusion

INTERVENTIONS:
Procedure: Kidney transplantation with MSCs infusion — Patients in Group A will receive the first MSCs infusion intravenously within 24 hours after kidney transplant operation , and the second infusion of MSCs will be performed two weeks later.
  Other Names: MSCs induction plus a standard or a lower dose of CNI
  Arms: A; B
Procedure: kidney transplantation without MSC infusion — kidney transplantation with standard immunosuppressive treatment regime
  Other Names: Anti-IL2R induction therapy with standard dose of CNI
  Arms: C

SUMMARY:
The goal of this study is to evaluate autologous MSCs as an alternative for antibody induction therapy in renal transplantation.

DETAILED DESCRIPTION:
Renal transplantation is the most common and successful type of organ transplantation. Induction therapy with antibody plus the maintenance immunosuppressive agents have greatly improved graft survival in renal transplantation. Since mesenchymal stem cells(MSCs)have been used successfully to treat graft versus host disease and show immune modulation function both in vitro and in vivo and may help in repairing damaged tissue(s), we evaluate autologous MSCs as an alternative for antibody induction therapy. Moreover, we examine if MSCs could improve the recovery of early function in transplanted kidney.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be between the ages of 18 and 60 years and meet the institution's criteria for renal transplantation for end-stage renal failure
* Patient is receiving the first renal transplant
* Patient is receiving a renal transplant only
* Women who are of child bearing potential must have a negative pregnancy test (urine test is acceptable) and agree to use reliable contraception for 1 year following transplant
* Willing to comply with the study visits
* Be able to sign informed consent document.

Note: The subjects do not need to be local residents in order to be eligible for this trial, but must be willing to reside in the area, or within a four hour drive, for the first three months of the protocol so that we can monitor them closely in the early post transplant period.

Exclusion Criteria:

* Previously received or is receiving an organ transplant other than a kidney
* Significant liver disease, defined as having continuously elevated AST (SGOT) or ALT (SGPT) levels greater than 3 times the upper value of the normal range within 28 days prior to study entry
* HIV infection.
* Surface antigen positive for HBV.
* Antibody positive for hepatitis C virus
* Recipient or donor is positive for tuberculosis (TB), under treatment for suspected TB, or previously exposed to TB
* Currently receiving an investigational drug or received an investigational drug within 30 days prior to transplant.
* Currently receiving any immunosuppressive agent.
* Clinically active bacterial, fungal, viral or parasitic infection
* Evidence for immunologic memory against donor.
* Recipients need antibody induction treatment before the operation.
* Current cancer or a history of cancer within the 5 years prior to study entry.
* Serious heart and lung diseases.
* Patients who's RPR is positive
* Pregnancy or breastfeeding.
* Have no ability to communicate.
* Any form of substance abuse, psychiatric disorder, or other condition that, in opinion of the investigator, may interfere with the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 165 (Actual)
Dates: Start 2008-03; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Incidence rate of biopsy-proven acute rejection and early renal function recovery | At 1 year post-transplant

SECONDARY OUTCOMES:
Patient and graft survival and prevalence of adverse events | At 1 year post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Jianming Tan, M.D and Ph.D, Study Director — Fuzhou General Hospital
Locations (1):
- Stem cell therapy center,Fuzhou General Hospital, Fuzhou, Fujian, China

REFERENCES:
- [Derived] Tan J, Wu W, Xu X, Liao L, Zheng F, Messinger S, Sun X, Chen J, Yang S, Cai J, Gao X, Pileggi A, Ricordi C. Induction therapy with autologous mesenchymal stem cells in living-related kidney transplants: a randomized controlled trial. JAMA. 2012 Mar 21;307(11):1169-77. doi: 10.1001/jama.2012.316. PMID 22436957